CLINICAL TRIAL: NCT00276744
Title: A Feasibility Study for Individualized Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: Individualized Drug Treatment for Treating Patients With Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because there was no longer an active laboratory component to this study.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0507; P30CA006973 (NIH); CDR0000455000; 05-04-14-02 (Other: JHM IRB)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Capecitabine; Docetaxel; Erlotinib Hydrochloride; Gemcitabine; Irinotecan; Mitomycin; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): PART A: Participants will have their tumors collected at the time of conventional surgery. Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Patients will then proceed to receive adjuvant treatment based on physician discretion and will be followed until disease progression.
  Capecitabine 1,5 mmol/kg Oral gavage 1- 5 days x 2 weeks Cetuximab 500 mg IP Twice a week x 2 weeks Docetaxel 20 mg/kg IV Once at week x 4 weeks Erlotinib 75 mg/kg IP 1-5 days x 2 weeks Gemcitabine 100 mg/kg IP Twice a week x 4 weeks Irinotecan 50 mg/kg IV Twice a week Mitomycin C 5 mg/kg IP One dose Rapamycin 4 mg/kg IP 1-5 days x 2 weeks
  PART B: At the time of progression, patients will be evaluated for Part B of the study and treated with the drug selected in Part A as the most active using approved doses and schedules of administration.
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: docetaxel; Drug: Erlotinib; Drug: Gemcitabine; Drug: Irinotecan; Drug: mitomycin C; Drug: rapamycin; Procedure: conventional surgery

INTERVENTIONS:
Biological: cetuximab — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
Drug: capecitabine — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: xeloda
Drug: docetaxel — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: taxotere
Drug: Erlotinib — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: tarceva
Drug: Gemcitabine — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: gemzar
Drug: Irinotecan — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: campto
Drug: mitomycin C — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: mitomycin
Drug: rapamycin — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.
  Other Names: sirolimus
Procedure: conventional surgery — Tumors will be implanted in nude mice and treated with a set of 8 commercially available anticancer drugs. Drugs will be ranked based in their activity from most to least active. Biological studies will be conducted in tumor tissues to better understand the response to tested drugs.

SUMMARY:
RATIONALE: Treating tumor tissue in the laboratory with different drugs may help doctors find the best drug for treating individual patients with pancreatic cancer.

PURPOSE: This phase II trial is studying an individualized drug treatment selection process, based on laboratory results, for treating patients with pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish tumor xenografts from patients with resectable adenocarcinoma of the pancreas who undergo surgical resection at Johns Hopkins Hospital.
* Determine the activity of a series of 10 anticancer drugs against these tumors in ex vivo studies.
* Determine the response rate, time to treatment failure, and 6-month survival rate in patients whose tumors were xenografted and treated in the mouse when treated with the most active agent identified in that model.
* Define determinants of susceptibility and resistance to the drugs in xenografted tumors.

OUTLINE:

* Part I (surgical resection, tumor xenografts generation, and drug selection): Patients undergo surgical resection. The resected tumor tissue is implanted in laboratory mice to generate tumor xenografts. The mice are then treated with a series of 10 approved anticancer drugs, whose anticancer activity are ranked from the most to the least effective based on response of the tumor xenografts. The most effective drug is identified for the individual patient. Patients for whom no drug is found to be effective are removed from the study. Patients who develop progressive disease after surgical resection and after mice data is available proceed to part II.
* Part II (individual patient treatment): Patients receive the most effective drug identified in part I in the absence of disease progression or unacceptable toxicity. The drugs may include bortezomib, capecitabine, cetuximab, docetaxel, erlotinib hydrochloride, gemcitabine hydrochloride, irinotecan hydrochloride, mitomycin C, sirolimus, or thalidomide.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
Part A

Inclusion Criteria

1. Suspected adenocarcinoma of the pancreas with resectable disease schedule to have surgical resection at the Johns Hopkins Hospital.
2. Age ≥ 18 years old.
3. Ability to understand and willingness to sign a written informed consent document.

Part B

Inclusion Criteria

1. Participation in Part A of the study with informative mouse xenograft data.
2. Histologically or cytologically confirmed diagnosis of invasive adenocarcinoma of the pancreas and peripancreatic adenocarcinoma, including distal cholangiocarcinoma, duodenal carcinoma, and ampullary pancreatic not amenable to curative treatment.
3. ECOG performance status 0 or 1
4. Age ≥ 18 years old.
5. Expected survival > 12 weeks.
6. No prior treatment for recurrent disease.
7. Willingness of male and female subjects, who are not surgically sterile or postmenopausal, to use reliable methods of birth control (oral contraceptives, intrauterine devices, or barrier methods used with a spermicide) for the duration of the study and for 30 days after the last dose of test article.
8. Adequate liver, renal and bone marrow functions.

WBC > 3,500 cells/mm3 ANC > 1,500 cells/mm3 Platelets > 100,000 cells/mm3 Hemoglobin ≥ 9 g/dl Serum creatinine 2 mg/dl Bilirubin 2 mg/dL ALT, AST, and alkaline phosphatase 5 times the upper limit of normal

Exclusion criteria

1. Patients in whom histologic or cytologic diagnosis is not consistent with adenocarcinoma.
2. Patients in whom histologic or cytologic diagnosis is consistent with non epithelial origin tumors, including adenosquamous, islet cell, cystadenoma or cystadenocarcinoma, carcinoid, small or large cell carcinoma, sarcoma, lymphoma and melanoma
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

4. Patients who have had any previous surgery, excluding minor procedures, dental work, skin biopsy, etc. within 4 weeks of enrollment.

5. Uncontrolled medical conditions that could potentially increase the risk of toxicities or complications when treated with chemotherapy. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.

6. Active infections.

7. History of another neoplasm except for non-metastatic, nonmelanoma skin cancers, < 5 years prior to enrollment.

8. Unable to provide informed consent.

9. Treatment with chemotherapy within 30 days of day 1 treatment.

10. Any unresolved chronic toxicity greater than CTCAE grade 2 from previous anticancer therapy (except alopecia).

11. Pregnant women are excluded from this study because the effects of the chemotherapy agents to be tested on the developing fetus are not known. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MMC, breast feeding should be discontinued if the mother is treated with the drug.

12. Patients must not have documented history of clinically significant cardiovascular disease including myocardial infarction (within 12 months prior to randomization), unstable angina, grade II or greater peripheral vascular disease, uncontrolled congestive heart failure or uncontrolled hypertension (SBP>170, DBP>95).

13. Patients with non informative xenograft data including patients whose tumors do not take in the mice, who progress before mice data is available or whose tumors do not respond to any of the selected agents.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2005-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Laheru, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villarroel MC, Rajeshkumar NV, Garrido-Laguna I, De Jesus-Acosta A, Jones S, Maitra A, Hruban RH, Eshleman JR, Klein A, Laheru D, Donehower R, Hidalgo M. Personalizing cancer treatment in the age of global genomic analyses: PALB2 gene mutations and the response to DNA damaging agents in pancreatic cancer. Mol Cancer Ther. 2011 Jan;10(1):3-8. doi: 10.1158/1535-7163.MCT-10-0893. Epub 2010 Dec 6. PMID 21135251

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 249 participants were enrolled however 240 received intervention in the study. Reason unknown and data is not accessible for the 9 remaining participants who were not assigned to intervention
Period: PART A
Arm/Group | Arm 1
Started | 240
Completed | 142
Not Completed | 98
Not completed — Reason unknown | 98
Period: PART B
Arm/Group | Arm 1
Started | 0 (This study was terminated before participants could reach this stage of the study.)
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated before participants could be entered into Part B.
Arm/Group | Arm 1
Number analyzed (Participants) | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 187
  >=65 years | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 125
Region of Enrollment [Number; unit: participants]
  United States | 240

OUTCOME MEASURES:

1. Primary Outcome: 6-month Overall Survival
Description: Percentage of patients survived at 6 months for patients whose tumors were xenografted and treated in the mouse when treated with the most active agent identified in that model
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 236
percentage of participants | 53

ADVERSE EVENTS:
Description: The patients all received FDA approved chemotherapy depending on the results in their mice, so adverse events were not monitored or assessed. Therefore adverse event data was not collected.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No